CLINICAL TRIAL: NCT04573595
Title: Fresenius Noninvasive Blood Pressure Validation - Three Phase Study PR 2020-377
Brief Title: Fresenius Noninvasive Blood Pressure Validation
Acronym: BPM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2020-377
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to provide supporting documentation for Noninvasive blood pressure measurement accuracy claims for Fresenius 5008S BPM Module and Cuffs on the intended population(s). The same arm sequential method with dual observer auscultation will be used to collect data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Blood Pressure Measurement — The purpose of this study is to provide supporting documentation for Noninvasive blood pressure measurement accuracy claims for Fresenius 5008S BPM Module and Cuffs on the intended population(s). The same arm sequential method with dual observer auscultation will be used to collect data.

SUMMARY:
The purpose of this study to collect blood pressure measurement values from the blood pressure measurement device on the Fresenius machine as compared to the standard method.

DETAILED DESCRIPTION:
This study is a comparative, single-center, non-randomized comparative study. After IRB approval, the study will be conducted in three Phases. The Fresenius 5008S BPM Module and Cuffs will be evaluated on a minimum of 120 subjects. Three reports will be generated and submitted to different regulatory bodies with the following minimum subject demographics:

* Phase 1: The submission to the United States Food and Drug Administration will include 85 adult and adolescents ages 13 and older.
* Phase 2: The submission to European agencies will contain 50 adult and adolescents ages 13 and older and 35 pediatric subjects ages 3-12.
* Phase 3: The submission to the China Food and Drug Administration will contain 73 adult and adolescents ages 13 and older and 12 pediatric subjects ages 3-12.

Each subject test is expected to take up to 1 hour. Data collection is expected to take 3-6 weeks for Phase 1. Phase 2 and 3 are expected to take an additional 2-4 weeks.

The Auscultator will have a normal audiogram before the study begins. All experimenters will review the protocol prior to test.

Testing will be conducted under normal office environment conditions.

Each subject or their legally authorized representative will be provided an IRB approved Informed Consent. Additionally, subject ages 7 to 17 years, a discussion about the study will be conducted to complete the Assent process for their participation. As applicable, subjects / authorized representatives will be told about any new information that might change their decision to participate. Representatives / subjects who have completed the informed consent and health questionnaire form and meet inclusion/exclusion criteria will be enrolled in the study if they meet desired blood pressure demographics. For Phase 3, an attempt will be made to enroll a person of Chinese origin in each of the cuffs used in the study.

Two trained observers will listen to the Korotkoff sounds at the brachial artery of the arm. The reference blood pressure measurements by the observers will be performed sequentially with the Device Under Test. The Device Under Test memory will be cleared prior to the next determination. In some cases, this may mean powering down the device to clear the previous readings.

The blood pressure measurements will be such that a reference measurement will be alternated with the Device Under Test measurement. The auscultator will wait a minimum of 60 seconds between each blood pressure determination. Each observer's recording of observations of the reference sphygmomanometer shall not be visible to the other observer. The observers will record the exact measurement heard during auscultation and will not round the blood pressure readings. The readings of the Device Under Test shall not be visible to either of these observers.

The observers will complete 1 or 2 initial baseline blood pressure measurements and then 3 to 8 NIBP measurements to be collected for the Accuracy evaluation.

* For Phase 1 and 2, any pair of observers' determinations with a difference greater than 4 mmHg shall be excluded per ANSI/AAMI/ISO 81060-2:2018.
* For Phase 3, any pair of observers' determinations with a difference greater than 10 mmHg shall be excluded and 90% of the observers' determinations shall be within 5 mmHg per YY 0670-2008.

If any determinations are excluded, additional pair(s) of determinations shall be taken to ensure that the needed number of valid test-reference pairs is available (up to a maximum of 8 paired readings) A minimum of 3 valid paired NIBP measurements are needed for the Accuracy analysis. Each subject test is expected to take up to 60 minutes for the enrollment / data collection process.

There are no deviations expected from this investigation plan, should deviations be needed, discussions will be conducted with the sponsoring company, Principal investigator and the IRB will be notified.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide an informed consent or have legally authorized representative consent to participate.
* Subject must be willing and able to comply with the study procedures.
* Subjects must be ≥ 13 years of age for Phase 1.
* Subjects must be ≥ 3 years of age for Phase 2 and 3.
* Subjects that are between 7 and 17 years of age must provide Assent to participate in the study.
* Subject or legally authorized representative must be able to read or write in English.
* Subjects must have an arm circumference in the range of 13-55cm or a thigh circumference in the range of 50-70 cm circumference.
* At least 30% of subjects shall be male and at least 30% of subjects shall be female.

Exclusion Criteria:

* Lack of Informed Consent
* Subjects with deformities or abnormalities that may prevent proper application of the Device Under Test.
* Subject is evaluated by the investigator or clinician and found to be medically unsuitable for participation in this study.
* Subjects with known heart dysrhythmias.
* Subjects with compromised circulation or peripheral vascular disease.
* Subjects with clotting disorders or taking blood thinners.
* Subjects that cannot tolerate sitting for up to 1 hour.
* Subject with a blood pressure demographic that has already been filled.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Validation of Blood Pressure Module (BPM) and Cuffs on the Fresenius Hemodialysis Machine | Baseline Comparator
  The Fresenius 5008S BPM with cuffs will be compared to the Reference sphygmomanometer via dual auscultator method. This will be a one-time measurement only no patient follow-up will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Arthure Cabrera, MD, Principal Investigator — Avista Adventist Hosptial, Staff Anesthesiologist
Locations (1):
- Clinimark, Site ID#001, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No